CLINICAL TRIAL: NCT01923311
Title: A Phase 2/3 Multicenter, Open-Label, Multicohort, Two-Part Study Evaluating the Pharmacokinetics (PK), Safety, and Antiviral Activity of Elvitegravir (EVG) Administered With a Background-Regimen (BR) Containing a Ritonavir-Boosted Protease Inhibitor (PI/r) in HIV-1 Infected, Antiretroviral Treatment-Experienced Pediatric Subjects
Brief Title: Two Part Study to Evaluate Pharmacokinetics, Safety, and Antiviral Activity of Elvitegravir Administered With a PI/r Background Regimen for ARV Treatment-Experienced Pediatric Participants
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-183-0160; 2013-001969-16 (EudraCT Number)
Record Dates: First submitted 2013-08-09; First posted 2013-08-15 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Acquired Immune Deficiency Syndrome (AIDS); HIV Infections
Keywords: Pediatrics; Adolescents; HIV; HIV-1; Treatment-experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — elvitegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (12 to < 18 years of age) (Experimental): Part A: No participants will be enrolled in Part A, as PK data is currently available for this age group.
  Part B: Participants will receive EVG plus a background regimen that includes a PI/r for up to 48 weeks. After Week 48, participants will be given the option to continue EVG therapy until the participant turns 18 and EVG is available for use in adults in the country in which the participant is enrolled, or the age appropriate EVG formulation becomes available for use in the country in which the participant is enrolled, or Gilead Sciences elects to terminate development of EVG in the applicable country.
  Interventions: Drug: EVG; Drug: Background regimen
- Cohort 2 (6 to < 12 years of age) (Experimental): Part A: Participants with HIV-1 RNA < 50 copies/mL will receive EVG plus a background regimen that includes a PI/r for 10 days. Participants with HIV-1 RNA > 1,000 copies/mL will receive EVG along with a newly constructed background regimen that includes a Pl/r for 48 weeks. Participants with HIV-1 RNA > 1,000 copies/mL can continue after Week 48.
  Part B: Following confirmation of exposure to EVG and based on safety and PK data assessed in Part A, participants will receive EVG plus a background regimen that includes a PI/r for up to 48 weeks. Participants who complete the 48-week follow-up in both Part A and Part B will be given the option to continue EVG therapy until the participant turns 18 and EVG is available for use in adults in the country in which the participant is enrolled, or the age appropriate EVG formulation becomes available for use in the country in which the participant is enrolled, or Gilead Sciences elects to terminate development of EVG in the applicable country.
  Interventions: Drug: EVG; Drug: Background regimen
- Cohort 3 (2 to < 6 years of age) (Experimental): Part A: Participants with HIV-1 RNA < 50 copies/mL will receive EVG plus a background regimen that includes a PI/r for 10 days.
  Part B: Following confirmation of exposure to EVG and based on safety and PK data assessed in Part A, participants will receive EVG plus a background regimen that includes a PI/r for up to 48 weeks. After Week 48, participants will be given the option to continue EVG therapy until the participant turns 18 and EVG is available for use in adults in the country in which the participant is enrolled, or the age appropriate EVG formulation becomes available for use in the country in which the participant is enrolled, or Gilead Sciences elects to terminate development of EVG in the applicable country.
  Interventions: Drug: EVG; Drug: Background regimen
- Cohort 4 (4 weeks to < 2 years of age) (Experimental): Part A: Participants with HIV-1 RNA < 50 copies/mL will receive EVG plus a background regimen that includes a PI/r for 10 days.
  Part B: Following confirmation of exposure to EVG and based on safety and PK data assessed in Part A, participants will receive EVG plus a background regimen that includes a PI/r for up to 48 weeks. After Week 48, participants will be given the option to continue EVG therapy until the participant turns 18 and EVG is available for use in adults in the country in which the participant is enrolled, or the age appropriate EVG formulation becomes available for use in the country in which the participant is enrolled, or Gilead Sciences elects to terminate development of EVG in the applicable country.
  Interventions: Drug: EVG; Drug: Background regimen

INTERVENTIONS:
Drug: EVG — Tablet (s) or tablet (s) for oral suspension (if unable to swallow) will be administered orally once daily
  Other Names: Vitekta®
Drug: Background regimen — Background regimen may consist of the following ritonavir (RTV)-boosted PIs (PI/r): lopinavir/r (Kaletra), atazanavir/r, darunavir/r, tipranavir/r, or fosamprenavir/r. For participants < 2 months old, only lopinavir/r is allowed. Use of additional antiretrovirals in background therapy may be allowed.

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability and steady-state PK and confirm the dose of EVG/r in HIV-1 infected, antiretroviral treatment-experienced children 4 weeks to <18 years of age.

The study consists of 2 parts: Part A and Part B. Part A will enroll participants with suppressed viremia (HIV-1 RNA < 50 copies/mL) or failing a current antiretroviral (ARV) regimen (HIV-1 RNA > 1,000 copies/mL only for participants in Cohort 2, Part A) to evaluate the steady state PK and confirm the dose of EVG. Part B will enroll participants who are failing a current ARV regimen (HIV-1 RNA > 1,000 copies/mL) to evaluate the safety, tolerability, and antiviral activity of EVG. The study consists of 4 age cohorts with each cohort including 2 parts (Part A and Part B) with the exception of the adolescent age cohort (Cohort 1: 12 to < 18 years old) containing Part B only.

ELIGIBILITY:
Key Inclusion Criteria:

Individuals must meet all of the following inclusion criteria to be eligible for participation in this study. Individuals with screening results that do not meet eligibility criteria will not be allowed to rescreen.

* HIV-1 infected male and female individuals 4 weeks (gestational age of at least 44 weeks) to less than 18 years of age at Baseline.
* Individuals are able to provide written assent if they have the ability to read and write.
* Parent or legal guardian able to provide written informed consent prior to any screening evaluations and willing to comply with study requirements.
* Body weight at screening greater than 5kg, 10.6kg, or 15kg dependent upon age cohort
* Adequate renal function
* Adequate hematologic function
* Hepatic transaminases (AST and ALT) less than or equal to 5 x upper limit of normal (ULN)
* Total bilirubin less than or equal to 1.5 mg/dL, or normal direct bilirubin
* Negative serum pregnancy test
* Individuals with evidence of suppressed viremia
* Individuals failing a current antiretroviral regimen at study entry
* Male and female individuals of childbearing potential must agree to utilize highly effective contraception methods while on study treatment or agree to abstain from heterosexual intercourse of reproductive potential throughout the study period and for 30 days following the last dose of study drug
* Must be willing and able to comply with all study requirements.

Key Exclusion Criteria:

Participants who meet any of the following exclusion criteria are not to be enrolled in this study.

* Individuals with CD4+ cell counts at Screening of less than 50, 75, or 200 cells/mm3 dependent on age cohort
* An AIDS defining condition with onset within 30 days prior to screening
* Life expectancy of less than 1 year
* For Individuals with HIV-1 RNA greater than 1,000 copies/mL at screening, prior treatment of any duration with an integrase strand transfer inhibitor.
* An ongoing serious infection requiring systemic antibiotic therapy at the time of screening.
* Evidence of active pulmonary or extra-pulmonary tuberculosis disease
* Anticipated requirement for rifamycin treatment while participating in the study.
* Have any serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with Individual's treatment, assessment, or compliance with the protocol.
* Individuals experiencing decompensated cirrhosis
* A history of or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma.
* Pregnant or lactating females.
* Current alcohol or substance abuse judged by the Investigator to potentially interfere with individual's compliance.
* Have history of significant drug sensitivity or drug allergy.
* Known hypersensitivity to the study drug, the metabolites, or formulation excipients.
* Have previously participated in an investigational trial involving administration of any investigational agent within 30 days prior to the study dosing.
* Participation in any other clinical trial without prior approval from sponsor is prohibited while participating in this trial.
* Individuals receiving ongoing therapy with any medication that is not to be taken with EVG or a component of the BR, including drugs not to be used with ritonavir

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 4 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2013-08-26 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (11):
- United States (3):
  - University of Colorado Denver, Aurora, Colorado
  - Duke University Medical Center, Durham, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- Universita degli Studi di Pavia - Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
- South Africa (2):
  - Be Part Yoluntu Centre, Cape Town
  - Rahima Moosa Mother and Child Hopsital, Johannesburg
- Spain (2):
  - Hospital Universitario De Getafe, Getafe, Madrid
  - Hospital 12 de Octubre, Madrid
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (HIV-NAT), Bangkok
  - Siriraj Hospital, Bangkok
- Joint Clinical Research Centre, Kampala, Uganda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, Asia, and Africa. The first participant was screened on 26 August 2013. The last study visit occurred on 03 November 2017.
Pre-assignment Details: 48 participants were screened.
  The study was discontinued after enrollment of only Cohort 1, Part B and Cohort 2, Part A. The study close-out was triggered by the voluntary withdrawal of single-agent Vitekta® sale based solely on low utilization of the product, and was not a result of any ongoing or new safety issue.
Groups:
- Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL: Elvitegravir (EVG) 50 mg, or 85 mg, or 150 mg tablet administered once daily (QD) for at least 48 weeks, based on body weight and dependent on the coadministered background regimen. (Background regimen may consist of the following ritonavir (RTV) boosted-protease inhibitors (PI/r): lopinavir/r (Kaletra; LPV/r), atazanavir/r (ATV/r), darunavir/r (DRV/r), tipranavir/r (TPV/r), or fosamprenavir/r (FPV/r). Use of additional antiretrovirals in background therapy was allowed.). After Week 48, participants were given the opportunity to continue receiving EVG in an extension phase, during which they attended study visits every 12 weeks, until they reached 18 years of age and EVG was commercially available for use in adults in the country in which they were enrolled; the age-appropriate EVG formulation became commercially available in the country in which they were enrolled; or Gilead elected to terminate the development of EVG.
- Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL: EVG 50 mg, or 85 mg tablet administered QD for 10 days, based on body weight and dependent on the coadministered background regimen. (Background regimen may consist of the following PI/r: LPV/r, ATV/r, DRV/r, TPV/r, or FPV/r. Use of additional antiretrovirals in background therapy was allowed.).
Period: Overall Study
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Started | 17 | 14
Completed | 0 | 13
Not Completed | 17 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Investigator's Discretion | 1 | 0
Not completed — Non-Compliance with Study Drug | 2 | 1
Not completed — Withdrew Consent | 1 | 0
Not completed — Study Terminated by Sponsor | 12 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who were enrolled into the study and received at least 1 dose of study drug.
Groups:
- Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL: EVG 50 mg, or 85 mg, or 150 mg tablet administered QD for at least 48 weeks with the option to continue receiving EVG after Week 48 in the extension phase, based on body weight and dependent on the coadministered background regimen. (Background regimen may consist of the following PI/r: LPV/r, ATV/r, DRV/r, TPV/r, or FPV/r. Use of additional antiretrovirals in background therapy was allowed.). After Week 48, participants were given the opportunity to continue receiving EVG in an extension phase, during which they attended study visits every 12 weeks, until they reached 18 years of age and EVG was commercially available for use in adults in the country in which they were enrolled; the age-appropriate EVG formulation became commercially available in the country in which they were enrolled; or Gilead elected to terminate the development of EVG.
- Total: Total of all reporting groups
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (2.9) | 9 (2.2) | 12 (3.8)
Age, Customized [Count of Participants; unit: Participants]
  Age 6 to < 12 Years | 2 | 14 | 16
  Age 12 to < 18 Years | 15 | 0 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 6 | 8 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 2 | 7
  Black | 11 | 10 | 21
  White | 0 | 2 | 2
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 17 | 13 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 7 | 8
  Italy | 1 | 0 | 1
  South Africa | 7 | 0 | 7
  Uganda | 3 | 3 | 6
  Thailand | 5 | 2 | 7
  Spain | 0 | 2 | 2
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.21 (0.802) | 1.33 (0.204) | 2.91 (1.576)
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 0 | 13 | 13
  ≥ 50 to ≤ 1000 copies/mL | 3 | 1 | 4
  > 1000 to ≤ 100000 copies/mL | 13 | 0 | 13
  > 100000 copies/mL | 1 | 0 | 1
Cluster of differentiation (CD4) Cell Count [Mean (Standard Deviation); unit: cells/uL] | 356.6 (249.45) | 810.8 (303.29) | 561.7 (354.74)
Cluster of differentiation (CD4) Cell Count Category [Count of Participants; unit: Participants]
  < 50 cells/uL | 0 | 0 | 0
  ≥ 50 to < 200 cells/uL | 6 | 1 | 7
  ≥ 200 to < 350 cells/uL | 3 | 0 | 3
  ≥ 350 to < 500 cells/uL | 4 | 0 | 4
  ≥ 500 cells/uL | 4 | 13 | 17
Cluster of differentiation (CD4) Percentage [Mean (Standard Deviation); unit: percentage (%)] | 17.8 (9.60) | 35.5 (9.11) | 25.8 (12.85)
Type of PI in Background Regimen (Excluding Ritonavir) [Count of Participants; unit: Participants]
  atazanavir | 8 | 1 | 9
  darunavir | 3 | 0 | 3
  lopinavir | 6 | 13 | 19

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of EVG
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Predose and up to 12 hours postdose on Day 10
Population: Intensive PK Analysis Set(EVG): all enrolled participants who received at least 1 dose of study drug and for whom steady-state pharmacokinetic profiles of the analyte of interest at the Intensive PK(Day 10) visit were evaluable.Includes 12 participants with screening HIV-1 RNA<50 copies/mL and 2 participants with screening HIV-1 RNA>1000 copies/mL.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Age 6 to < 12 Years: PK results were summarized for all participants age 6 to < 12 years as one group.
  EVG 50 mg, or 85 mg tablet administered QD for 10 days (participants with screening HIV-1 RNA < 50 copies/mL), or at least 48 weeks (participants with screening HIV-1 RNA > 1000 copies/mL), based on body weight and dependent on the coadministered background regimen (For participants receiving ATV/r or LPV/r, the EVG dose was 50 mg for participants ≥ 17 to < 30 kg and 85 mg for participants ≥ 30 kg).
Arm/Group | Age 6 to < 12 Years
Number analyzed (Participants) | 14
h*ng/mL | 24028.3 (7302.44)
Statistical Analysis 1: Comparison: Age 6 to < 12 Years; To determine whether the proposed EVG dose in children achieved similar systemic exposure to adults, statistical comparisons were performed with PK data from the current study (test) and adult data from population PK modeling in study GS-US-183-0145 (NCT00708162) (reference); Test type: Equivalence — A total of 12 test study participants compared to 334 HIV-infected reference study participants will provide at least 90% power to conclude exposure equivalence of EVG AUCtau in test study vs reference study, assuming the expected geometric mean ratio is 1, equivalency boundary is 70% to 143%, 2 one-sided tests are each performed at an alpha level of 0.05, and the standard deviation of EVG AUCtau is 0.36 ng•h/mL (natural log scale, estimated from EVG population PK modeling); GLSM Ratio (%) (Test/Reference) = 135.73, 90% CI 2-sided [116.24 to 158.49]

2. Primary Outcome: Pharmacokinetic (PK) Parameter: Cmax of EVG at Day 10
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Predose and up to 12 hours postdose on Day 10
Population: Intensive PK Analysis Set (EVG)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Age 6 to < 12 Years
Number analyzed (Participants) | 14
ng/mL | 2022.1 (599.94)
Statistical Analysis 1: Comparison: Age 6 to < 12 Years; To determine whether the proposed EVG dose in children achieves similar systemic exposure to adults, statistical comparisons were performed with PK data from the current study (test) and adult data from population PK modeling in study GS-US-183-0145 (NCT00708162) (reference); Test type: Equivalence — A total of 12 test study participants compared to 334 HIV-infected reference study participants will provide at least 90% power to conclude exposure equivalence of EVG Cmax in test study vs reference study, assuming the expected geometric mean ratio is 1, equivalency boundary is 70% to 143%, 2 one-sided tests are each performed at an alpha level of 0.05, and the standard deviation of EVG Cmax is 0.28 ng•h/mL (natural log scale, estimated from EVG population PK modeling); GLSM Ratio (%) (Test/Reference) = 146.68, 90% CI 2-sided [127.35 to 168.94]

3. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events
Time Frame: Baseline up to the last dose date plus 30 days (maximum exposure: 173.6 weeks for participants age 6 to < 18 Years Screening HIV-1 RNA > 1000 copies/mL and 2.0 weeks for participants age 6 to < 12 Years Screening HIV-1 RNA < 50 copies/mL)
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL: EVG 50 mg, or 85 mg, or 150 mg tablet administered QD for at least 48 weeks, based on body weight and dependent on the coadministered background regimen. (Background regimen may consist of the following PI/r: LPV/r, ATV/r, DRV/r, TPV/r, or FPV/r. Use of additional antiretrovirals in background therapy was allowed.). After Week 48, participants were given the opportunity to continue receiving EVG in an extension phase, during which they attended study visits every 12 weeks, until they reached 18 years of age and EVG was commercially available for use in adults in the country in which they were enrolled; the age-appropriate EVG formulation became commercially available in the country in which they were enrolled; or Gilead elected to terminate the development of EVG.
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 17 | 14
percentage of participants | 100.0 | 35.7

4. Primary Outcome: Percentage of Participants Experiencing Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each subject. The criteria used to grade laboratory results were as follows: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), and Grade 4 (life-threatening).
Time Frame: as for outcome 3
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 17 | 14
percentage of participants
  Grade 1 | 11.8 | 50.0
  Grade 2 | 35.3 | 21.4
  Grade 3 | 35.3 | 7.1
  Grade 4 | 17.6 | 0

5. Secondary Outcome: Pharmacokinetic (PK) Parameter: Ctau of EVG
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Predose and up to 12 hours postdose on Day 10
Population: Intensive PK Analysis Set (EVG)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Age 6 to < 12 Years
Number analyzed (Participants) | 14
ng/mL | 494.3 (261.05)

6. Secondary Outcome: Pharmacokinetic (PK) Parameter: CL/F of EVG
Description: CL/F is defined as the apparent oral clearance following administration of the drug.
Time Frame: Predose and up to 12 hours postdose on Day 10
Population: Intensive PK Analysis set (EVG)
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Age 6 to < 12 Years
Number analyzed (Participants) | 14
mL/h | 2863.5 (871.07)

7. Secondary Outcome: Pharmacokinetic (PK) Parameter: Vz/F of EVG
Description: Vz/F is defined as the apparent volume of distribution of the drug.
Time Frame: Predose and up to 12 hours postdose on Day 10
Population: Participants in the Intensive PK Analysis Set: EVG with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Age 6 to < 12 Years
Number analyzed (Participants) | 13
mL | 39508.3 (14071.51)

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 as Defined by the FDA Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Full Analysis Set: all participants who were enrolled in the study and received at least 1 dose of study drug. Participants in the Full Analysis Set with available data were analyzed. Week 24 HIV-1 RNA copies for participants with screening HIV-1 RNA < 50 copies/mL were not analyzed due to the short duration of treatment (10 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 17 | 0
percentage of participants | 76.5 [50.1 to 93.2] |

9. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the FDA Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with available data were analyzed. Week 48 HIV-1 RNA copies for participants with screening HIV-1 RNA < 50 copies/mL were not analyzed due to the short duration of treatment (10 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 17 | 0
percentage of participants | 58.8 [32.9 to 81.6] |

10. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 24 as Defined by the FDA Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 400 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed. Week 24 HIV-1 RNA copies for participants with screening HIV-1 RNA < 50 copies/mL were not analyzed due to the short duration of treatment (10 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 17 | 0
percentage of participants | 82.4 [56.6 to 96.2] |

11. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 48 as Defined by the FDA Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 400 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 17 | 0
percentage of participants | 76.5 [50.1 to 93.2] |

12. Secondary Outcome: Change From Baseline in Plasma Log₁₀ HIV-1 RNA at Week 24
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed. Week 24 Plasma Log₁₀ HIV-1 RNA data for participants with screening HIV-1 RNA < 50 copies/mL was not analyzed due to the short duration of treatment (10 days).
Measure: Mean (Standard Deviation); unit: Log₁₀ copies/mL
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 16 | 0
Log₁₀ copies/mL | -2.44 (1.132) |

13. Secondary Outcome: Change From Baseline in Plasma Log₁₀ HIV-1 RNA at Week 48
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set with available data were analyzed. Week 48 Plasma Log₁₀ HIV-1 RNA data for participants with screening HIV-1 RNA < 50 copies/mL was not analyzed due to the short duration of treatment (10 days).
Measure: Mean (Standard Deviation); unit: Log₁₀ copies/ mL
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 15 | 0
Log₁₀ copies/ mL | -2.23 (1.293) |

14. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 24
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed. Week 24 CD4 Cell Count data for participants with screening HIV-1 RNA < 50 copies/mL was not analyzed due to the short duration of treatment (10 days).
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 16 | 0
cells/uL | 77.6 (138.06) |

15. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set with available data were analyzed. Week 48 CD4 Cell Count data for participants with screening HIV-1 RNA < 50 copies/mL was not analyzed due to the short duration of treatment (10 days).
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 15 | 0
cells/uL | 131.3 (195.04) |

16. Secondary Outcome: Change From Baseline in CD4 Percentage at Week 24
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed. Week 24 CD4 percentage data for participants with screening HIV-1 RNA < 50 copies/mL group was not analyzed due to the short duration of treatment (10 days).
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 16 | 0
percentage (%) | 3.56 (4.109) |

17. Secondary Outcome: Change From Baseline in CD4 Percentage at Week 48
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set with available data were analyzed. Week 48 CD4 percentage data for participants with screening HIV-1 RNA < 50 copies/mL group was not analyzed due to the short duration of treatment (10 days).
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 15 | 0
percentage (%) | 5.31 (5.772) |

18. Secondary Outcome: Tanner Stage Evaluation by Sex at Week 24
Description: Tanner Stage (pubic hair and breasts for females; pubic hair and genitalia for males) at Week 24 visit was summarized using frequency count and percentage. Tanner Stages is a scale that defines physical measurements of development based on external primary and secondary sex characteristics. It was used in this study to assess pubertal development with values ranging from Stage 1 (pre-pubertal characteristics) to Stage 5 (adult or mature characteristics).
Time Frame: Week 24
Population: Participants in the Safety Analysis Set with available data were analyzed. Tanner Stage Assessments were not defined for participants with screening HIV-1 RNA < 50 copies/mL because there were no postbaseline assessments scheduled in the protocol for these participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 17 | 0
Participants
  Female: Pubic Hair: number analyzed (Participants) | 11 | 0
  Female: Pubic Hair: Stage 1 | 1 |
  Female: Pubic Hair: Stage 2 | 0 |
  Female: Pubic Hair: Stage 3 | 4 |
  Female: Pubic Hair: Stage 4 | 5 |
  Female: Pubic Hair: Stage 5 | 1 |
  Female: Pubic Hair: Missing | 0 |
  Female: Breasts: number analyzed (Participants) | 11 | 0
  Female: Breasts: Stage 1 | 0 |
  Female: Breasts: Stage 2 | 0 |
  Female: Breasts: Stage 3 | 3 |
  Female: Breasts: Stage 4 | 5 |
  Female: Breasts: Stage 5 | 3 |
  Female: Breasts: Missing | 0 |
  Male: Pubic Hair: number analyzed (Participants) | 6 | 0
  Male: Pubic Hair: Stage 1 | 2 |
  Male: Pubic Hair: Stage 2 | 2 |
  Male: Pubic Hair: Stage 3 | 0 |
  Male: Pubic Hair: Stage 4 | 0 |
  Male: Pubic Hair: Stage 5 | 2 |
  Male: Pubic Hair: Missing | 0 |
  Male: Genitalia: number analyzed (Participants) | 6 | 0
  Male: Genitalia: Stage 1 | 2 |
  Male: Genitalia: Stage 2 | 2 |
  Male: Genitalia: Stage 3 | 0 |
  Male: Genitalia: Stage 4 | 0 |
  Male: Genitalia: Stage 5 | 2 |
  Male: Genitalia: Missing | 0 |

19. Secondary Outcome: Tanner Stage Evaluation by Sex at Week 48
Description: Tanner Stage (pubic hair and breasts for females; pubic hair and genitalia for males) at Week 48 visit was summarized using frequency count and percentage. Tanner Stages is a scale that defines physical measurements of development based on external primary and secondary sex characteristics. It was used in this study to assess pubertal development with values ranging from Stage 1 (pre-pubertal characteristics) to Stage 5 (adult or mature characteristics).
Time Frame: Week 48
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 17 | 0
Participants
  Female: Pubic Hair: number analyzed (Participants) | 11 | 0
  Female: Pubic Hair: Stage 1 | 0 |
  Female: Pubic Hair: Stage 2 | 1 |
  Female: Pubic Hair: Stage 3 | 4 |
  Female: Pubic Hair: Stage 4 | 4 |
  Female: Pubic Hair: Stage 5 | 1 |
  Female: Pubic Hair: Missing | 1 |
  Female: Breasts: number analyzed (Participants) | 11 | 0
  Female: Breasts: Stage 1 | 0 |
  Female: Breasts: Stage 2 | 0 |
  Female: Breasts: Stage 3 | 2 |
  Female: Breasts: Stage 4 | 5 |
  Female: Breasts: Stage 5 | 3 |
  Female: Breasts: Missing | 1 |
  Male: Pubic Hair: number analyzed (Participants) | 6 | 0
  Male: Pubic Hair: Stage 1 | 3 |
  Male: Pubic Hair: Stage 2 | 1 |
  Male: Pubic Hair: Stage 3 | 0 |
  Male: Pubic Hair: Stage 4 | 1 |
  Male: Pubic Hair: Stage 5 | 1 |
  Male: Pubic Hair: Missing | 0 |
  Male: Genitalia: number analyzed (Participants) | 6 | 0
  Male: Genitalia: Stage 1 | 2 |
  Male: Genitalia: Stage 2 | 2 |
  Male: Genitalia: Stage 3 | 0 |
  Male: Genitalia: Stage 4 | 0 |
  Male: Genitalia: Stage 5 | 2 |
  Male: Genitalia: Missing | 0 |

20. Secondary Outcome: Age of First Menses
Description: Age of first menses for female participants.
Time Frame: Baseline through end of study (maximum exposure: 173.6 weeks for participants age 6 to < 18 Years with Screening HIV-1 RNA > 1000 copies/mL and 2.0 weeks for participants age 6 to < 12 Years with Screening HIV-1 RNA < 50 copies/mL)
Population: Participants in the Safety Analysis Set with available data were analyzed. Age of First Menses for participants ages 6 to < 12 years with screening HIV-1 RNA < 50 copies/mL was not analyzed because none of the participants reached their first menstruation cycle during or prior to the study.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 11 | 0
years | 13 (1.9) |

21. Secondary Outcome: Palatability of Oral Suspension Formulation of EVG in Appropriate Age Group
Time Frame: Up to Week 48
Population: Palatability was only to be assessed for participants taking EVG suspension formulation. As no participants were dosed with the EVG oral suspension formulation, no data are available on its palatability.
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Adherence to EVG
Description: Adherence was calculated as the number of pills taken divided by number of pills prescribed multiplied by 100.
Time Frame: Baseline up to the last dose date (maximum exposure: 173.6 weeks for participants age 6 to < 18 Years Screening HIV-1 RNA > 1000 copies/mL and 2.0 weeks for participants age 6 to < 12 Years Screening HIV-1 RNA < 50 copies/mL)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of pills
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
Number analyzed (Participants) | 17 | 14
percentage of pills | 91.1 (8.94) | 100.0 (0.00)

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (maximum exposure: 173.6 weeks for participants age 6 to < 18 Years Screening HIV-1 RNA > 1000 copies/mL and 2.0 weeks for participants age 6 to < 12 Years Screening HIV-1 RNA < 50 copies/mL)
Description: Safety Analysis Set: all participants who were enrolled and received at least 1 dose of study drug.
Arm/Group | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/14
Other Adverse Events (participants affected / at risk) | 17/17 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL (N=17) | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL (N=14)
Bronchitis (Infections and infestations) | 1 | 0
Plasmodium falciparum infection (Infections and infestations) | 0 | 1
Skin candida (Infections and infestations) | 1 | 0
Syphilis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Age 6 to < 18 Years With Screening HIV-1 RNA > 1000 Copies/mL (N=17) | Age 6 to < 12 Years With Screening HIV-1 RNA < 50 Copies/mL (N=14)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 3 | 0
Dental caries (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 2 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0
Body tinea (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 2 | 0
Parotid abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Varicella (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Crystal urine present (Investigations) | 1 | 0
Lymph node palpable (Investigations) | 1 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 0
Parosmia (Nervous system disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Genital ulceration (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2013-04-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT01923311/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT01923311/SAP_001.pdf